CLINICAL TRIAL: NCT04327830
Title: Decision-making Needs of Older Adults Receiving Home Care From the Perspective of Older Adults, Their Caregivers and Inter-disciplinary Health and Social Care Providers: Participatory Mixed Methods Study
Brief Title: What Older Adults and Their Caregivers Need for Making Better Decisions at Home
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: St Elizabeth Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: MCD315
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Aging
Keywords: Shared decision making; Home care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older adults and their caregivers: Older adults who have received or are receiving home care services and their caregivers
  Interventions: Other: Decisional needs assessment
- Interdisciplinary health and social care providers: Interdisciplinary health and social care providers who provide home care services to older adults
  Interventions: Other: Decisional needs assessment

INTERVENTIONS:
Other: Decisional needs assessment — Assessment of decision-making needs

SUMMARY:
Most Canadians wish to stay at home in their old age. As older adults stay at home with the support of home and community services, they are often faced with difficult decisions, such as "Who will look after me when I can't look after myself any more, or if I have dementia?" or "Should I move to a nursing home, or stay here?" Care providers in the home and community can support older adults and their families make these difficult decisions by providing them with information they need and asking them about their values and preferences. By helping older adults and their families know more about their choices and choose options that reflect what is important to them, care providers can work with their clients to help them make informed health decisions together. In this fellowship, the investigators will study what supports are needed for older adults to make informed health decisions from the perspective of older adults, caregivers and front-line care providers in the home and community setting across Canada. This can help improve the home and community services provided to older adults (and their caregivers) so that older adults (and their caregivers) can make better decisions together with their health care team.

DETAILED DESCRIPTION:
Introduction Shared decision making is an interpersonal process whereby healthcare providers collaborate with and support patients in decision-making. Older adults receiving home care need support with decision-making (e.g., information on risks and benefits of options). This study will explore what older adults and their caregivers need for making better health-related decisions at home, and what health and social care providers need for supporting their home care clients with decision-making.

Methods and analysis This two-phase sequential exploratory mixed methods study will be conducted in a pan-Canadian healthcare organization, St Elizabeth Health Care. First, the investigators will create a participant advisory group (one older adult, one caregiver and two care providers) to advise us throughout the research process. In Phase 1 (qualitative), the investigators will recruit a convenient sample of older adults and caregivers receiving home care to participate in open-ended semi-structured interviews to discuss what health-related decisions they face at home and what they need for making better decisions (e.g. types of knowledge, sources of support). In Phase 2 (quantitative), interdisciplinary health and social care providers (e.g., nurses, personal support workers, occupational therapists, physiotherapists) will be invited to answer an online survey to share their views on the decision-making needs of older adults and their caregivers. The survey will include close-ended questions informed by findings from the qualitative interviews in Phase 1. Finally, qualitative and quantitative results will be triangulated from the perspective of older adults, caregivers and health and social care providers. Results will be reported using EQUATOR guidelines.

ELIGIBILITY:
Inclusion Criteria:

* older adults who have received, or are receiving home care services
* caregivers of older adults who have received, or are receiving home care services
* interdisciplinary health and social care providers who provide home care services for older adults

Exclusion Criteria:

* no experience receiving or providing home care services

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Older adults who have received or are receive home care services (and their caregivers)
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Decision making needs of older adults who receive home care services and their caregivers. | About 60 minutes
  Interview of older adults and their caregivers. Open-ended questions guide by the Ottawa Decision Support Framework (ODSF).
What health and social care providers need to support older adults and their caregivers with making decisions. | 5 to 10 minutes
  Survey of interdisciplinary health and social care providers, based on the Ottawa Decision Support Framework (ODSF) factors contributing to difficulty.

SECONDARY OUTCOMES:
-Health and social care providers opinion how often older adults faced difficult decisions. -Shared decision-making. -Others participants involved in the decision making. | 5 to 10 minutes
  * Opinion frequency; 5-point Likert scale always to never.
  * Shared decision-making generic approach in 5 questions; 5-point Likert scale always to never.

CONTACTS AND LOCATIONS:
Overall Officials: France Legare, Study Chair — Laval University /SE Health
Locations (1):
- CERSSPL, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Statistics Canada. Home health care and related services [Report on the Internet]. Ottawa: Statitics Canada, 2017 (cited July 31, 2019). Accessed on Feb 10, 2020 from: https://www150.statcan.gc.ca/n1/daily-quotidien/190731/dq190731c-eng.htm
- [Background] 2. Canadian Institute for Health Information. Home care expenditures in the NHEX Database [Technical note on the Internet] Ottawa: The Institute; 2017 (cited November 2017). Accessed on Feb 20, 2020 from: https://www.cihi.ca/sites/default/files/document/technical_notes_on_home_care-nhex2017-en.pdf.
- [Derived] Lai C, Holyoke P, Plourde KV, Decary S, Legare F. What older adults and their caregivers need for making better health-related decisions at home: a participatory mixed methods protocol. BMJ Open. 2020 Nov 9;10(11):e039102. doi: 10.1136/bmjopen-2020-039102. PMID 33168556